CLINICAL TRIAL: NCT06297837
Title: Adaptive Prediction of Antimicrobial Susceptibility and Its Implementation to Improve the Management of Urinary Tract Infection
Brief Title: ADAPT-AST (Adaptive Antimicrobial Susceptibility Testing)
Acronym: ADAPT-AST
Status: Active, not recruiting | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: LHS0205
Record Dates: First submitted 2024-02-08; First posted 2024-03-07 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-11

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to improve the way urinary tract infections (UTIs) are tested for antibiotic resistance. The main questions it aims to answer are:

* Can the investigators use a method called Bayesian causal inference to create or check clinical prediction models that help predict if certain antibiotics will work for a urinary infection, using patient information from the National Health Service (NHS)?
* Can this new ADAPT-AST method, which uses data and a smarter approach, do a better job of testing for urinary infection than the old methods? Will it help doctors make quicker decisions and save resources by being more efficient?

Participants in this study will not be receiving treatments. The study will involve:

Using statistical methods to predict UTI test results based on patient data. Evaluating whether this new approach can provide doctors with more timely and useful information for treating UTIs.

Assessing whether it can help save money and resources in the lab and pharmacy.

DETAILED DESCRIPTION:
The aim of this study is to develop and evaluate an adaptive informatics approach for laboratory antimicrobial susceptibility testing (AST) for urinary tract infection (UTI) pathogens compared with current practice to improve patient outcomes, reduce AMR risks and reduce waste of laboratory resources.

UTI is a leading cause of community and hospital acquired infection and a major driver of antimicrobial prescribing in primary and secondary care. The continued proliferation of AMR also increasingly limits treatment choices for many UTIs. Despite the importance of UTI, antimicrobial susceptibility testing (AST) of urine specimens is based on inflexible 'one-size-fits' all standard operating procedures (SOPs). Either a very large unfocused panel of antimicrobials is immediately tested (leading to wasted resources), or more commonly, and particularly in low or middle income (LMIC) settings, a selected subset of antimicrobials is tested at day one prior to a second or even third panel of antimicrobials. Such an approach does not adapt to prior information such as previous resistance patterns, antimicrobial prescribing, or demographic information, despite these factors being powerful (strong) predictors of resistance. This results in imprecise, inefficient, and inequitable provision of antimicrobial susceptibility information, which provides suboptimal support of decisions for treatment of UTI.

This project will use statistical techniques based on Bayesian causal inference to predict urine AST results and prioritise testing using patient demographics, prescribing, admission, and microbiology laboratory care data. The clinical utility of resulting algorithms will be evaluated in terms of their ability to increase the number, timeliness and appropriateness of usable AST results available to clinicians, and their ability to reduce laboratory resource costs through better test prioritisation. The anticipated benefits of a successfully developed, evaluated, and implemented system are faster and more precise treatments of UTI in patients with drug-resistant organisms and more efficient resource management, particularly in laboratory and pharmacy workflows.

ELIGIBILITY:
Inclusion Criteria:

* o The specimens for which AST predictions & recommendations will be made are urine specimens processed by LCL Microbiology laboratory taken from patients ≥ 18 years old in LUHFT and/or GP locations that grew organisms within the period of the study dataset; these are the only specimens for which AST results will be available to train and test ADAPT-AST. Predictions will be made for all urine specimen types, including mid-stream urines, catheter specimens of urine and nephrostomy urine.

Exclusion Criteria:

* Urine specimens processed by LCL that did not grow organisms within the period of the study dataset
* Urine specimens taken from patients < 18 years old
* Predictions will be made for asymptomatic bacteriuria screening specimens in pregnant women who have had specimens sent from a GP, but not those which have been sent from Liverpool Womens' NHS Foundation Trust (LWfT) Predictions for non-bacterial organisms grown in urine (i.e., fungi) will not be made.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a suspected Urinary Tract Infection
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
The overall number of susceptible results per panel available at day 1 | 2 years
  The overall number of susceptible results per panel available at day 1

SECONDARY OUTCOMES:
The number of susceptible results per panel available for WHO AWaRe Access category agents at day 1 | 2 years
  The number of susceptible results per panel available for WHO AWaRe Access category agents at day 1
The number of susceptible results per panel for orally-administrable agents available at day 1 | 2 years
  The number of susceptible results per panel for orally-administrable agents available at day 1
The number of susceptible results per panel for intravenously-administrable agents available at day 1 | 2 years
  The number of susceptible results per panel for intravenously-administrable agents available at day 1
The proportion of panels with no results available for WHO AWaRe Access category agents at day 1 | 2 years
  The proportion of panels with no results available for WHO AWaRe Access category agents at day 1
The proportion of panels with no susceptible results of any kind available at day 1 | 2 years
  The proportion of panels with no susceptible results of any kind available at day 1
The proportion of WHO Access agent susceptible results for the agent with the highest utility value | 2 years
  The proportion of WHO Access agent susceptible results for the agent with the highest utility value
The proportion of susceptible results of any kind for the agent with the highest utility value | 2 years
  The proportion of susceptible results of any kind for the agent with the highest utility value

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, North West, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/37/NCT06297837/Prot_ICF_000.pdf